CLINICAL TRIAL: NCT01549509
Title: A Phase I Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 Recombinant Adenovirus-5 Vector Vaccine, VRC-HIVADV014-00-VP Administered Alone or Administered as a Boost to a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA009-00-VP, in Uninfected Adult Volunteers in Uganda
Brief Title: Evaluating the Safety of and Immune Response to an HIV Vaccine in Healthy, HIV-Uninfected Adults in Uganda
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RV 156A; 10469 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VRC-HIVADV014-00-VP Vaccine (Experimental): All participants will receive one injection of the study vaccine (VRC-HIVADV014-00-VP) in their upper arm at study entry.
  Interventions: Biological: VRC-HIVADV014-00-VP Vaccine

INTERVENTIONS:
Biological: VRC-HIVADV014-00-VP Vaccine — All participants will receive one injection in their upper arm of 1 x 10^10 particle units (PU)/mL of VRC-HIVADV014-00-VP at study entry.

SUMMARY:
The RV 156A clinical trial is evaluating an experimental HIV vaccine in people who are not infected with HIV. Participants in that study are randomly assigned to receive either the HIV vaccine or placebo. This study will enroll people who are participating in the RV 156 study. In this study, researchers will evaluate the safety of and immune response to a different experimental HIV vaccine in people who participated in the RV 156 study.

DETAILED DESCRIPTION:
RV 156A is a single site, phase 1 open label study with accrual restricted to participants in RV 156. Participants in the RV 156 study were randomly assigned to receive three injections of either placebo or the VRC-HIVDNA009-00-VP vaccine. All participants in this study will receive one injection of a different experimental HIV vaccine, VRC-HIVADV014-00-VP. The purpose of this study is to evaluate the safety and immunogenicity of the VRC-HIVADV014-00-VP vaccine in people who participated in the RV 156 study. Researchers will examine the differences in the immune response to the VRC-HIVADV014-00-VP vaccine between people who received placebo in the RV 156 study and people who received the VRC-HIVDNA009-00-VP vaccine in the RV 156 study.

A projected number of up to 29 volunteers will be enrolled from the Makerere University site in Uganda. At study entry, all participants will undergo a physical examination, medical history review, vital sign measurements, and blood and urine collection. They will also receive counseling for HIV prevention and pregnancy prevention. Participants will then receive one injection of the VRC-HIVADV014-00-VP vaccine in their upper arm. They will remain in the clinic for 30 to 45 minutes for observation and monitoring. For 3 days after the vaccination, participants will record their temperature and any adverse symptoms in a diary. Additional study visits will occur at Days 3, 14, 28, 42, 84, 168, 252, and 336. At each visit, participants will undergo the same study procedures that they completed at the study entry visit.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 40 years old at the time of RV 156 enrollment
* Available for follow-up for the duration of the study (13 months)
* Satisfactory completion of an Assessment of Understanding prior to enrollment, defined as 90% correct with three opportunities to take the test
* Able and willing to sign the informed consent form
* Willing to receive HIV counseling and testing in accordance with Ugandan Ministry of Health guidelines
* Willing to not engage in high-risk behavior for HIV infection during the study as defined by the protocol and amenable to risk-reduction counseling and discussion of HIV infection risks
* In good general health
* Physical examination and laboratory results without clinically significant findings within 45 days prior to rAd5 boost injection
* Have participated in RV 156 and received all three required vaccinations

Laboratory Criteria within 45 days prior to enrollment:

* Hemoglobin greater than 11.0 g/dL for women and 12.5 g/dL for men or accompanied by site physician approval and above the site's lower limit of normal (LLN) range
* White blood cell count (WBC) of 3,300 to 12,000 cells/mm^3 (in the absence of clinical or pathological etiology)
* Absolute neutrophil count (ANC) within the institutional normal ranges and greater than or equal to 1,000 cells/mm^3 or accompanied by site physician approval
* Total lymphocyte count greater than 800 cells/mm^3
* Platelets equal to 125,000 to 550,000 cells/mm^3
* Alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) less than 1.25 times the upper limit of normal (ULN)
* Serum creatinine less than 1.0 times the ULN range
* Normal urinalysis, defined as dipstick with negative glucose, negative or trace protein, and negative or trace hemoglobin (blood) or determined to be not clinically significant by site principal investigator
* Negative serology for HIV infection (e.g., enzyme linked immunosorbent assay [ELISA] test, western blot [WB]) and HIV ribonucleic acid (RNA) below detection limits of Food and Drug Administration (FDA)-approved viral load diagnostic assay

Pregnancy-Specific Criteria:

* Negative serum-human chorionic gonadotropin (HCG) pregnancy test for all women. A female participant must meet one of the following criteria from the screening visit and throughout the duration of the study:

  1. No reproductive potential because of a hysterectomy, bilateral oophorectomy, or tubal ligation. Documentation from qualified medical doctor must be obtained for confirmation of procedure. OR
  2. Participant agrees to consistently practice contraception at least 21 days prior to vaccination and throughout the duration of the study (13 months).
* More information on this criterion can be found in the protocol

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during the period of study participation
* Immunosuppressive or cytotoxic medications within the past 6 months with the exception of corticosteroid nasal spray for allergic rhinitis or topical corticosteroids for an acute uncomplicated dermatitis
* Blood products within 120 days prior to HIV screening
* Immunoglobulin within 60 days prior to HIV screening
* Live attenuated vaccines within 30 days prior to initial study vaccine administration
* Investigational research agents within 30 days prior to initial study vaccine administration
* Medically indicated subunit or killed vaccines, e.g., influenza, pneumococcal, or allergy treatment with antigen injections, within 14 days of study vaccine administration
* Current anti-tuberculosis (TB) prophylaxis or therapy

People with a history of any of the following clinically significant conditions will be excluded:

* Serious adverse reactions to vaccines such as anaphylaxis, hives, respiratory difficulty, angioedema, or abdominal pain
* Autoimmune disease or immunodeficiency
* Asthma that is unstable or required emergent care, urgent care, hospitalization, or intubation during the past 2 years. Asthma that has required the use of oral or intravenous corticosteroids during the past 2 years.
* Diabetes mellitus (type I or II), with the exception of gestational diabetes
* Thyroid disease, including history of thyroidectomy and diagnoses that required medication within the past 36 months
* Serious angioedema episodes within the previous 36 months or requiring medication in the previous 2 years
* Hypertension that is not well controlled by medication or blood pressure greater than or equal to 150/100 mm Hg (either or both values) at second screening and/or entry visits
* Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with intramuscular (IM) injections or blood draws
* Active syphilis documented by exam or serology unless positive serology is because of remote treated infection or positive rapid plasma regain/venereal disease research laboratory (RPR/VDRL) test is not associated with positive Treponemal specific serology
* Malignancy that is active, treated malignancy for which there is not reasonable assurance of sustained cure, or malignancy that is likely to recur during the period of the study
* Seizure disorder other than febrile seizures under the age of 2
* Asplenia or splenic hypoplasia (complete or partial lack of splenic function) or any condition resulting in the absence of a functional spleen or removal of the spleen
* Psychiatric condition that precludes compliance with the protocol, past or present psychoses, past or present bipolar disorder, or suicidal attempts
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to protocol adherence or a person's ability to give informed consent

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Local reactogenicity signs and symptoms | Measured through Day 336
Systemic reactogenicity signs and symptoms | Measured through Day 336
Laboratory measures of safety | Measured through Day 336
Adverse and serious adverse experiences | Measured through Day 336

CONTACTS AND LOCATIONS:
Overall Officials: Fred Wabwire-Mangen, MBChB, PhD, Principal Investigator — Makerere University Walter Reed Project
Locations (1):
- Makerere University Walter Reed Project (MUWRP), Kampala, Uganda